CLINICAL TRIAL: NCT07237113
Title: Effects of Omega-3 Fatty Acid Supplementation on Muscle Damage and Oxylipin Production Induced by Eccentric Exercise in Young Men
Brief Title: Muscle Recovery After Omega-3 Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencias de la Salud, Universidad de O'Higgins (Other)
Collaborators: Universidad Nacional Andres Bello (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, Sebastian Jannas-Vela, Associate Professor, Instituto de Ciencias de la Salud, Universidad de O'Higgins
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 020/2021
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2021-08

CONDITIONS: Damage Muscle
Keywords: omega-3; oxylipins; exercise-induced muscle damage; specialized pro-resolving mediators

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a double-blind manner to two supplementation groups: (a) placebo (yellow maltodextrin) or (b) omega-3 (EPA and DHA). Prior to the start of the supplementation period, participants will undergo venous blood sampling, indirect markers of muscle damage testing, oxygen consumption testing, and the eccentric exercise protocol on one leg (6 sets of 10 repetitions at 80% of 1 repetition maximum). Immediately after, 1, 2, 24, 48, 72, and 96 hours after the eccentric exercise session, muscle damage will be assessed, and venous blood samples will be obtained. The following day, participants will begin their 8-week supplementation protocol with omega-3 or a placebo. After the supplementation period, participants will perform the same tests as at the beginning and will perform the eccentric exercise session on the opposite leg.
Who Masked: Participant, Investigator
Masking Description: The masking process will ensure that both the participants and the investigators involved in the study remain unaware of the treatment assignments throughout the entire duration of the study. A unique identification code will be assigned to each participant upon enrollment, which conceals their treatment allocation. The allocation sequence will be generated by a person not directly involved in the study. The capsules in the experimental intervention and the control treatment, will be packaged identically to maintain visual similarity. The packaging materials and labeling will be designed to be indistinguishable between the two groups. In addition, all outcome assessments and data collection procedures will be performed by personnel who are blinded to the treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control (Placebo Comparator): The participants will be supplemented with 5 capsules per day of a placebo-filled gelatin capsule.
  Interventions: Dietary Supplement: Placebo
- Omega-3 (Experimental): The participants will be supplemented with 5 capsules per day of Omega UP (Newscience, Chile) equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA.
  Interventions: Dietary Supplement: Omega

INTERVENTIONS:
Dietary Supplement: Placebo — The participants will be supplemented with 5 capsules per day of a placebo-filled gelatin capsule for 8 weeks.
  Arms: Placebo control
Dietary Supplement: Omega — The participants will be supplemented with 5 capsules per day of Omega UP (Newscience, Chile), equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA for 8 weeks
  Arms: Omega-3

SUMMARY:
In recent decades, omega-3 eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) have been proposed as potential therapeutic agents for minimizing muscle damage induced by eccentric exercise, especially when supplementation is long-term (> 6 weeks) and at high doses (> 1 g/d). However, no study has analyzed whether these effects are mediated by an increase in oxylipins (metabolites derived from EPA and DHA), which play an essential role in the muscle regeneration process. The objective of the present study is to determine the effect of eight weeks of high-dose omega-3 fatty acid supplementation on blood oxylipin levels and their association with muscle function and markers of muscle damage after high-intensity eccentric exercise in young men.

DETAILED DESCRIPTION:
Research question Does supplementation with high doses of omega-3 for eight weeks reduce muscle damage induced by a session of high-intensity eccentric exercise in young men? Is the response to eccentric exercise related to an increase in oxylipins derived from omega-3 fatty acids? Hypothesis Long-term supplementation (8 weeks) with high doses of omega-3 (3 g/d) will increase the concentration of oxylipins in the blood, which will be associated with less muscle damage after an eccentric exercise protocol in young men.

General objective To determine the effect of eight weeks of high-dose omega-3 fatty acid supplementation on blood oxylipin levels and indirect markers of muscle damage after high-intensity eccentric exercise in young men.

Specific objectives

1. To determine the effect of eight weeks of high-dose omega-3 fatty acid supplementation on blood oxylipin levels after high-intensity eccentric exercise in young men.
2. To determine the effect of eight weeks of high-dose omega-3 fatty acid supplementation on muscle function and markers of muscle damage after high-intensity eccentric exercise in young men.
3. Associate blood oxylipin levels with changes in muscle function and markers of muscle damage induced by a session of eccentric exercise, before and after high-dose omega-3 fatty acid supplementation in young men.

Methodology This study is an experimental, prospective, double-blind design. Sample size: The sample size calculation establishes a minimum of 12 subjects per group based on an α level of 0.05 and a power (1-β) of 0.8, assuming an estimated maximum strength loss difference of 22% after eccentric exercise (effect size = 1.06) between the omega-3 and control groups, based on a previous study (1). However, 15 participants will be recruited per group to account for a 20% dropout rate.

Methodology: Thirty young men will be recruited through posters and social media advertisements. Participants will be randomly assigned in a double-blind manner to two supplementation groups: (a) placebo (yellow maltodextrin) or (b) omega-3 (EPA and DHA). Prior to the start of the supplementation period, participants will undergo venous blood sampling, indirect markers of muscle damage testing, oxygen consumption testing, and the eccentric exercise protocol on one leg (6 sets of 10 repetitions at 80% of 1 repetition maximum). Immediately after, 1, 2, 24, 48, 72, and 96 hours after the eccentric exercise session, muscle damage will be assessed and venous blood samples will be obtained. The following day, participants will begin their 8-week supplementation protocol with omega-3 or placebo. After the supplementation period, participants will perform the same tests as at the beginning and will perform the eccentric exercise session on the opposite leg.

Exclusion criteria: Participants must not have performed regular strength training during the 6 months prior to the start of the study. Participants must also not be taking medications that affect inflammation or cardiovascular responses to exercise and must have a BMI of less than 30 kg/m2. Finally, participants must not consume fish more than twice a week and must not have taken any omega-3 supplements for three months prior to the study or be allergic to fish. Participants will be asked to have the Covid-19 vaccine. Participants will be fully informed about the nature and possible risks of the experimental procedures before providing their written informed consent approved by the Ethics Committee.

Supplementation: Participants will be supplemented with 5 capsules per day (5 g/d) of Omega Up OMEGA 3 (2.5 g/d of DHA and 0.5 g/d of EPA) or placebo. The dose used is in accordance with the recommendation of the EFSA (European Food Safety Authority), has been shown to be safe, incorporated into cell membranes, and to produce significant improvements in overall health (2,3).

Eccentric exercise protocol: The eccentric exercise protocol will consist of 6 sets of 10 repetitions of 45º leg presses performed at 80% of 1RM only in their eccentric phase, with 90 seconds of rest between sets performed on one leg (4). The concentric phase of the movement will be performed by one of the researchers.

Surveys: Two surveys will be conducted, the first on food consumption frequency, focused on quantifying the average intake of omega-3 fatty acids from the diet. Second, the validated IPAQ questionnaire will be used to quantify physical activity in participants (5).

Oxygen consumption test: Participants will perform an incremental test on a cycle ergometer (Lifecycle 9500HR; LifeFitness, Rosemont, IL, USA). Maximum power and VO2peak values will be obtained. The test will begin with 4 minutes at 50 W and will increase by 25 W every minute until exhaustion (6).

Maximum isometric strength (MVC): The MVC of the knee extensors of both legs will be measured at 90° of knee flexion on a quadriceps chair equipped with a load cell (Reverse S, USA). From this assessment, the rate of force development (RFD) will be calculated as a more sensitive marker of muscle stiffness and function.

Muscle pain: Thigh pain when sitting and standing from a chair 3 times will be assessed using a visual analog scale (100 cm), where 0 is no pain and 100 is maximum pain.

Thigh circumference: The exercised leg will be measured in the middle area. Measurements will be taken three times by the same examiner, and the average of these three measurements will be used for statistical analysis. A non-stretchable tape measure will be used. (Lufkin Executive Thinline, Maryland, USA)(7) Creatine kinase (CK) activity: 35uL will be extracted from the blood sample (below) and analyzed for CK activity in blood (Reflotron, Roche).

Blood samples: Venous blood samples will be obtained and immediately centrifuged to obtain plasma (1000 g for 10 minutes at 4°C) and erythrocyte fraction (3000 × g for 10 minutes at 20°C). Both fractions will be frozen at -80°C.

Phospholipid fatty acid composition (analysis of fatty acids in blood and GR): Quantitative extraction of total lipids from erythrocytes and plasma will be performed according to Bligh and Dyer (8) with the addition of BHT. Fatty acid methyl esters (FAME) from erythrocytes and plasma will be prepared according to Morrison and Smith (9). FAMEs will be extracted with 0.5 mL of hexane. FAMEs will be identified and quantified by gas-liquid chromatography on Agilent equipment (model 7890B, Santa Clara, CA, USA) equipped with a capillary column (Agilent HP-88, 100 m × 0.250 mm; ID 0.25 μm) and a flame ionization detector (FID). Identification and quantification of FAMEs will be achieved by comparing the retention times and peak area percentage values of unknown samples with those of the commercial lipid standard (Nu-Chek Prep Inc., Elysian, MN, USA). C23:0 will be used as the internal standard (Nu-Chek Prep Inc., Elysian, MN, USA). Data will be processed using the Hewlett-Packard Chemstation software system.

SPM analysis of plasma lipid mediators: Plasma samples (400 μL) will be analyzed in duplicate for oxylipins by HPLC/MS/MS as described previously (10). Briefly, deuterated internal standards (Cayman Chemicals) will be added to plasma samples and adjusted to pH <3.0 prior to solid-phase extraction using Strata-X-SPE columns (Phenomenex) preconditioned with methanol, followed by water at pH 3.0. Samples will be loaded onto the columns, washed, and free SPMs will be eluted with 100% methanol. The eluate will then be dried and resuspended in solvent A (water/acetonitrile/formic acid, 70/30/0.02 v/v/ v) for oxylipin analysis by HPLC/MS/MS, using a Luna 5-μm C18 column (100 Å, 250 × 2.0 mm, Phenomenex) on a Shimadzu Nexera XR HPLC, coupled to an ABSciex QTRAP 6500 MS operating in negative mode with electrospray ionization. Oxylipins will be eluted with the following gradient: 100% solvent A between 0 and 1 min, and then solvent B (acetonitrile/isopropyl alcohol, 50/50, v/v) is increased linearly to 25% at 3 min, 45% at 11 min, 60% at 13 min, 75% at 18 min, and 90% at 18.5 min. Solvent B is then held at 90% until 20 min, reduced to 0% at 21 min, and held until 25 min. Oxylipins will be quantified using the stable isotope dilution method.

Statistical analysis: Results will be expressed as mean ± standard deviation. Differences will be evaluated using a two-way analysis of variance (ANOVA) with Fisher's post hoc test (LSD) for multiple comparisons between groups and evaluation times. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants between 18 and 40 years

Exclusion Criteria:

* Participants must not have performed regular strength training during the 6 months prior to the start of the study.
* Participants must also not be taking medications that affect inflammation or cardiovascular responses to exercise and must have a BMI of less than 30 kg/m2.
* Participants must not consume fish more than twice a week and must not have taken any omega-3 supplements for three months prior to the study or be allergic to fish.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Maximum isometric voluntary contraction strength loss | Pre and post intervention (8 weeks)
  Change in MVC strength loss 0, 2, 24, 48, and 72 hours after.
Plasma oxylipins | Pre and post intervention (8 weeks)
  Levels of plasma oxylipins

SECONDARY OUTCOMES:
Peak aerobic capacity | Pre and post intervention (8 weeks)
  Incremental cycling test to exhaustion using a recumbent cycle ergometer to measure aerobic capacity.
Dietary assessment | Pre and post intervention (8 weeks)
  Dietary record over three days (two consecutive weekdays and one weekend day)
Fatty acid composition | Pre and post intervention (8 weeks)
  Quantitative extraction of total lipids from erythrocytes and plasma.
Thigh circumference | Pre and post intervention (8 weeks)
  The exercised leg will be measured in the middle area.
Creatine kinase | Pre and post intervention (8 weeks)
  Blood CK activity
Physical activity levels | Pre and post intervention (8 weeks)
  IPAQ questionnaire will be used to quantify physical activity in participants
Muscle soreness | Pre and post intervention (8 weeks)
  Thigh muscle soreness was quantified using a 100-mm visual analog scale (VAS) in which 0 indicated no pain and 100 represented the worst pain imaginable
Vertical Jump Performance | Pre and post intervention (8 weeks)
  Unilateral jump height will be measured with squat jump (SJ) and countermovement jumps (CMJ)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de O'Higgins, Rancagua, Libertador Bernardo O'Higgins, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Penailillo L, Blazevich A, Numazawa H, Nosaka K. Metabolic and muscle damage profiles of concentric versus repeated eccentric cycling. Med Sci Sports Exerc. 2013 Sep;45(9):1773-81. doi: 10.1249/MSS.0b013e31828f8a73. PMID 23475167
- [Result] Lv ZT, Zhang JM, Zhu WT. Omega-3 Polyunsaturated Fatty Acid Supplementation for Reducing Muscle Soreness after Eccentric Exercise: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Biomed Res Int. 2020 Apr 20;2020:8062017. doi: 10.1155/2020/8062017. eCollection 2020. PMID 32382573
- [Result] Levy BD, Clish CB, Schmidt B, Gronert K, Serhan CN. Lipid mediator class switching during acute inflammation: signals in resolution. Nat Immunol. 2001 Jul;2(7):612-9. doi: 10.1038/89759. PMID 11429545
- [Result] Gabbs M, Leng S, Devassy JG, Monirujjaman M, Aukema HM. Advances in Our Understanding of Oxylipins Derived from Dietary PUFAs. Adv Nutr. 2015 Sep 15;6(5):513-40. doi: 10.3945/an.114.007732. Print 2015 Sep. PMID 26374175
- [Result] Markworth JF, Maddipati KR, Cameron-Smith D. Emerging roles of pro-resolving lipid mediators in immunological and adaptive responses to exercise-induced muscle injury. Exerc Immunol Rev. 2016;22:110-34. PMID 26853678
- [Result] Tsuchiya Y, Yanagimoto K, Nakazato K, Hayamizu K, Ochi E. Eicosapentaenoic and docosahexaenoic acids-rich fish oil supplementation attenuates strength loss and limited joint range of motion after eccentric contractions: a randomized, double-blind, placebo-controlled, parallel-group trial. Eur J Appl Physiol. 2016 Jun;116(6):1179-88. doi: 10.1007/s00421-016-3373-3. Epub 2016 Apr 16. PMID 27085996
- [Result] Ramos-Campo DJ, Avila-Gandia V, Lopez-Roman FJ, Minarro J, Contreras C, Soto-Mendez F, Domingo Pedrol JC, Luque-Rubia AJ. Supplementation of Re-Esteri fi ed Docosahexaenoic and Eicosapentaenoic Acids Reduce Inflammatory and Muscle Damage Markers after Exercise in Endurance Athletes: A Randomized, Controlled Crossover Trial. Nutrients. 2020 Mar 9;12(3):719. doi: 10.3390/nu12030719. PMID 32182747
- [Result] Gerling CJ, Mukai K, Chabowski A, Heigenhauser GJF, Holloway GP, Spriet LL, Jannas-Vela S. Incorporation of Omega-3 Fatty Acids Into Human Skeletal Muscle Sarcolemmal and Mitochondrial Membranes Following 12 Weeks of Fish Oil Supplementation. Front Physiol. 2019 Mar 29;10:348. doi: 10.3389/fphys.2019.00348. eCollection 2019. PMID 30984028
- [Result] BLIGH EG, DYER WJ. A rapid method of total lipid extraction and purification. Can J Biochem Physiol. 1959 Aug;37(8):911-7. doi: 10.1139/o59-099. No abstract available. PMID 13671378
- [Result] MORRISON WR, SMITH LM. PREPARATION OF FATTY ACID METHYL ESTERS AND DIMETHYLACETALS FROM LIPIDS WITH BORON FLUORIDE--METHANOL. J Lipid Res. 1964 Oct;5:600-8. No abstract available. PMID 14221106
- [Result] Gabbs M, Zahradka P, Taylor CG, Aukema HM. Time Course and Sex Effects of alpha-Linolenic Acid-Rich and DHA-Rich Supplements on Human Plasma Oxylipins: A Randomized Double-Blind Crossover Trial. J Nutr. 2021 Mar 11;151(3):513-522. doi: 10.1093/jn/nxaa294. PMID 33097936